CLINICAL TRIAL: NCT06108284
Title: Impact of Negative Pressure Ventilation in Patients Hospitalized with Acute Hypercapnic Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Hayek Medical (Unknown)
Responsible Party: Principal Investigator, Dennis Chairman, Assistant Professor of Clinical Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2094467
Record Dates: First submitted 2023-10-09; First posted 2023-10-31 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: eligible patients will be randomized to either the conventional arm (non invasive positive pressure ventilation) vs the intervention arm using the Biphasic Cuirass Ventilation.
Masking Description: can't be done as the two devices are completely different.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional Arm (No Intervention): Patients will be placed on Non invasive positive pressure ventilation per current standard of care.
- Intervention Arm (Active Comparator): Patient in this arm will be placed on Biphasic Cuirass Ventilation
  Interventions: Device: Intervention Arm (Biphasic cuirass ventilation)

INTERVENTIONS:
Device: Intervention Arm (Biphasic cuirass ventilation) — Patients in this arm will be placed on Biphasic cuirass ventilation
  Arms: Intervention Arm

SUMMARY:
The study aims to find if using a Biphasic Cuirass Ventilation is as effective as using a Non invasive Positive Pressure Ventilation in patients admitted with acute hypercapnic respiratory failure.

DETAILED DESCRIPTION:
Patients presenting via Emergency Room or inpatients who are noted to be in acute hypercapnic respiratory failure will be approached for consent and if they are agreeable will be randomized to the standard of care arm which would be the use of Bilevel Positive pressure ventilation via face mask vs the intervention arm which would use the Biphasic Cuirass Ventilation.

Patients will be monitored and treated in the Medical ICU and will be regularly clinically assessed as per usual standard of care. The study investigators will obtain periodic Arterial/Venous Blood gas sampling to assess for improvement or lack thereof in patients Carbon dioxide levels.

If patients' condition doesn't improve or deteriorates their primary treating physician will have full authority to withdraw such patients from study and or change the modality of the patient's treatment.

This is a pilot study, and the investigators are aiming to compare the success rate of Biphasic cuirass ventilation when compared to non-invasive positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* admission diagnosis of hypercapnic respiratory failure
* pH between 7.20-7.35 in an ABG sample or pH between 7.16-.31 in a venous sample.

Exclusion Criteria:

* age <21
* Pregnant
* Inmate/Prisoner
* Contraindication for cuirass ventilator (open chest wound, flail chest, prior thoracic surgery)
* Chest wall defect, neuromuscular disease or diaphragmatic paralysis.
* BMI >50

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Resolution of Hypercapnic Respiratory Failure | 1-3 days
  Resolution of Hypercapnic Respiratory failure will be assessed and compared with the current standard of care which is non invasive positive pressure ventilation using Arterial or Venous Blood Gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chairman, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospitals, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data to anyone outside the study.

REFERENCES:
- [Background] Plant PK, Owen JL, Elliott MW. Early use of non-invasive ventilation for acute exacerbations of chronic obstructive pulmonary disease on general respiratory wards: a multicentre randomised controlled trial. Lancet. 2000 Jun 3;355(9219):1931-5. doi: 10.1016/s0140-6736(00)02323-0. PMID 10859037
- [Background] Dolmage TE, De Rosie JA, Avendano MA, Goldstein RS. Effect of external chest wall oscillation on gas exchange in healthy subjects. Chest. 1995 Feb;107(2):433-9. doi: 10.1378/chest.107.2.433. PMID 7842774